CLINICAL TRIAL: NCT01020097
Title: Is 18F-EF5 PET Imaging Useful in Determining the Prognosis of Newly Diagnosed Head and Neck Squamous Cell Carcinoma?
Brief Title: Fluorine F 18 EF5 Positron Emission Tomography in Assessing Hypoxia in Patients With Newly Diagnosed Stage I, Stage II, Stage III, or Stage IV Head or Neck Squamous Cell Cancer of the Oral Cavity, Oropharynx, and Larynx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 17308
Record Dates: First submitted 2009-11-18; First posted 2009-11-24 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Squamous Cell Carcinoma
Keywords: Stage 1 squamous cell carcinoma of the larynx
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Immunohistochemistry; Biopsy; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Other): Patients undergo fluorine F-18 EF5 positron emission tomography imaging. Scana are performed 180 minutes following injection.
  Interventions: Drug: fluorine F18 EF5; Procedure: immunohistochemistry staining method; Procedure: biopsy; Procedure: Positron Emission tomography

INTERVENTIONS:
Drug: fluorine F18 EF5 — Given IV
  Other Names: 18F-EF5
Procedure: immunohistochemistry staining method — Correlative study
  Other Names: immunohistochemistry
Procedure: biopsy — Correlative study
  Other Names: biopsies
Procedure: Positron Emission tomography — Undergo scan
  Other Names: FDG-PET, PET, PET scan, tomography, emission computed

SUMMARY:
Rationale: Diagnostic procedures, such as positron emission tomography, using the drug fluorine F 18-EF5 to find oxygen in tumor cells may help in planning cancer treatment.

Purpose: This clinical trial studies fluorine F 18-EF5 positron emission tomography in assessing hypoxia in patients with newly diagnosed stage I, stage II, stage III, or stage IV squamous cell cancer of the oral cavity, oropharynx, and larynx.

DETAILED DESCRIPTION:
Detailed DescriptionPRIMARY OBJECTIVES:

I. Describe the patterns and levels of 18F-EF5 in Stage 1 - 4 de novo HNSCC of the oral cavity, oropharynx and larynx.

II. Determine whether the 18F-EF5 PET images are predictive of patient outcome (event-free survival; EFS and overall survival; OS).

III. Determine whether any statistically significant prognostic relationships found in the corresponding grant are independent of nodal status.

SECONDARY OBJECTIVES:

I. Explore the relationship between 18F-EF5 signal and other measures of hypoxia (serum OPN; HIF1alpha protein expression), proliferation (Ki67+ cells/high power field (HPF)), apoptosis and radiation resistance (pAkt expression).

OUTLINE:

Patients undergo fluorine F 18-EF5 positron emission tomography imaging. Scans are performed 180 minutes following injection.

After completion of study, patients are followed at 2-4 weeks and 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed and/or clinical and imaging evidence of a Stage 1-4 de novo mass in the larynx, pharynx or oral cavity
* Treatment plan should include Surgery (Biopsy or Excision) and may be followed by radiation and/ or concurrent chemotherapy
* Patients' disease must not require emergency surgical attention
* The need for tracheotomy and/or feeding tube placement preceding definitive surgery is not a contradiction for participation
* Patients must have a Karnofsky performance status >= 70
* Patients must have a clinical condition and physiologic status for which the standard initial therapy is surgical biopsy or resection
* Patients must have normal organ and marrow function as defined below:
* WBC > 2,000/mm^3
* Platelets > 100,000/mm^3
* Total bilirubin
* Creatinine
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation (1 month)
* Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Serum pregnancy testing will be required for women of childbearing age
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* History of allergic reactions attributed to Flagyl (metronidazole), which has a chemical structure similar to EF5
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women and women who are breastfeeding
* Patients whose clinical status requires that surgery for their HNSCC be performed emergently or in a time course that does not allow scheduling of an 18F-EF5 PET scan preceding surgery and chemoradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
18F-EF5 standardized uptake values (SUV) | Study completion
  Data on 18F-EF5 signal are collected from multiple sections of the tumor via PET imaging. The outcomes of interest, are 18F-EF5 standardized uptake values (SUV) and/or tumor to normal tissue T:N ratios.
Tumor to normal tissue (T:N) ratios | Study completion
  Data on 18F-EF5 signal are collected from multiple sections of the tumor via PET imaging. The outcomes of interest, are 18F-EF5 standardized uptake values (SUV) and/or tumor to normal tissue T:N ratios.

SECONDARY OUTCOMES:
Event-free survival and overall survival | 5 years
  Length of time from end of treatment to recurrence or death

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States